CLINICAL TRIAL: NCT03782857
Title: Prevention After Stroke - a Nurse-led Physician-Supervised Model. A Feasibility Study
Brief Title: Prevention After Stroke - a Nurse-led Physician-supervised Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nete Hornnes (Other)
Responsible Party: Sponsor-Investigator, Nete Hornnes, Research Nurse, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-41-0429
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 to intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Initiation/stepwise escalation of antihypertensive medication in case of blood pressure above individual target Initiation/stepwise escalation of cholesterol lowering medication in case of LDL-cholesterol above individual target Advice on healthy lifestyle and life long adherence to preventive medication
  Interventions: Behavioral: Intervention
- Control group (No Intervention): Participants had the usual treatment: all patients were invited to one visit in the outpatient clinic three months after discharge with a diagnosis of stroke/TIA

INTERVENTIONS:
Behavioral: Intervention — Prevention of recurrent stroke, myocardial infarction and death Stepwise escalation of preventive medication Life style counselling including adherence to preventive treatment
  Arms: Intervention group

SUMMARY:
The study evaluates the effect of early follow up in a preventive clinic with stepwise treatment of high blood pressure and lowering blood cholesterol. Half the participants were randomized to the preventive clinic group and the other half to control group with the usual treatment: one visit to the outpatient clinic three months after discharge with a diagnosis of stroke or transient ischemic attack (TIA)

DETAILED DESCRIPTION:
Hypertension is the most important modifiable risk factor for recurrent stroke. Several studies have shown that less than 40% of stroke survivors are treated to target one year after stroke The investigator performed a feasibility study to test a model of treating this important risk factor in a hospital setting The investigator used a stepwise escalation of treatment of both blood pressure and blood cholesterol to individual targets according to patients' diagnosis of stroke, comorbidity and age

ELIGIBILITY:
Inclusion Criteria: Patients diagnosed with a stroke during stay in the stroke unit of Herlev Hospital

Exclusion Criteria: Severe stroke giving a modified Rankin Scale score >4, severe cognitive deficits or dementia, discharge to a nursing home

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2013-12-17 (Actual); Study Completion 2013-12-17 (Actual)

PRIMARY OUTCOMES:
Blood pressure treated to target | At follow up 10 months after inclusion in the study
  The investigator used individual targets of blood pressure: In case of hemorrhagic stroke: BP<130/80 mm Hg, in case of ischemic heart disease: BP target according to stroke diagnosis, but no lower than 130/80 mm Hg, in case of diabetes or chronic kidney disease: BP<130/80 mm Hg, age>80 years: <150/90 mm Hg, others: <140/90 mm Hg

SECONDARY OUTCOMES:
Reduction in blood pressure | At follow up 10 months after inclusion in the study
  Difference between blood pressure at inclusion in the study and blood pressure measured at final follow up

OTHER OUTCOMES:
Reduction in LDL-cholesterol | At follow up 10 months after inclusion in the study
  Difference between LDL-cholesterol at inclusion in the study and LDL-cholesterol measured at final follow up
LDL-cholesterol treated to target | At follow up 10 months after inclusion in the study
  In non-diabetic participants with ischemic stroke the target of lipid lowering treatment was LDL<2.5 mmol/l and <2.0 mmol/l in case of diabetes
Intensification of preventive treatment | From discharge from the stroke unit to final follow up in study
  Proportion of participants who had an intensification of antihypertensive / lipid lowering medication since discharge
Adherence with preventive medication | At follow up 10 months after inclusion in the study
  Proportion of participants with at least 80% adherence with preventive medication
Healthy lifestyle | At follow up 10 months after inclusion in the study
  Proportion of participants on a healthy diet, moderate physical activity for four hours/week, smoking cessation in baseline daily smokers, reduction of an overuse of alcohol to recommended level
Time to cardiovascular complications | From inclusion in the study to a median of 65 (61-66) months after inclusion
  Time to recurrent stroke, myocardial infarction and death in months

CONTACTS AND LOCATIONS:
Overall Officials: Nete Hornnes, MPH,Ph.d, Principal Investigator — Department of Neurology, Herlev Hospital, 2730 Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No